CLINICAL TRIAL: NCT04060004
Title: The Effects of Dry Needling on the Superficial Neck Musculature in Patients With Chronic Myofascial Pain: A Randomized Controlled Trial
Brief Title: The Effects of Dry Needling on the Superficial Neck Musculature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Ricardo Medrano de la Fuente, Physiotherapist, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.0 14/12/2018
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Neck Pain
Keywords: physical therapy
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Electric Stimulation Therapy; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Electrotherapy + therapeutic exercise
  Interventions: Other: Electrotherapy + therapeutic exercise
- Experimental group 1 (Experimental): Electrotherapy + therapeutic exercise + dry needling
  Interventions: Other: Dry needling; Other: Electrotherapy + therapeutic exercise
- Experimental group 2 (Placebo Comparator): Electrotherapy + therapeutic exercise + sham dry needling
  Interventions: Other: Sham dry needling; Other: Electrotherapy + therapeutic exercise

INTERVENTIONS:
Other: Dry needling — Dry needling is a technique used by physiotherapists.
  Arms: Experimental group 1
Other: Sham dry needling — Sham dry needling is a technique used by physiotherapists to compare the effects of dry needling.
  Arms: Experimental group 2
Other: Electrotherapy + therapeutic exercise — Standard care of neck pain.

SUMMARY:
The term myofascial pain refers to the existence of myofascial trigger points (MTP), which are defined as hypersensitive points in a tense band of skeletal muscle, which can cause referred pain or autonomous phenomena.

To address the treatment of myofascial trigger points, conservative and invasive techniques have been proposed. Dry needling is one of the invasive techniques that have been shown to be effective in improving pain and function in patients with myofascial trigger points.

This trial aims to analyse the effectiveness of dry needling in patients with myofascial neck pain.

DETAILED DESCRIPTION:
The main objective of the study is to analyze the effects of dry needling on the superficial neck musculature in patients with chronic myofascial neck pain in terms of pain, functional capacity, mobility, psychosocial variables and motor control compared with both sham dry needling group and control group.

In addition, a secondary objective is to analyze the relationships between the psychosocial variables and the results obtained in the variables analyzed in the patients belonging to the three groups.

For this purpose the investigators conduct a randomized controlled trial double-blind. Patients included are randomized into 3 groups. One receives dry needling, another one receives sham dry needling, and the last one is a control group.

The hypothesis of this study is that patients in the real dry needling group will improve more compared to patients in the sham dry needling group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myofascial neck pain
* Presence of at least one active myofascial trigger point on the superficial neck musculature
* Neck pain of at least 3 months
* Age 18-70
* Pain intensity between 20 and 100 mm in the Analog Visual Scale
* Neck disability index (NDI) greater than or equal to 15 points
* Spanish speakers
* Patients who do not present contraindications for the use of dry needling (anticoagulants, nickel allergy or belenophobia)
* Patients who have not received physiotherapy or pharmacological treatment for neck pain for the last three months

Exclusion Criteria:

* History of cervical trauma
* Cervical spine surgery
* Vertebral fracture
* Cervical pain associated with whiplash
* Red flags (tumor, metabolic disorders or rheumatoid arthritis)
* Inflammatory lesion in the neck region
* Pregnancy
* Fibromyalgia diagnosis
* Neck pain associated with radiculopathy
* Patients pending legal litigation
* Psychiatric pathology diagnosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Neck pain | Baseline.
  The investigators measure the neck pain with Visual Analogue Scale (VAS) at baseline.
Neck pain | Through study completion, an average of 11 days.
  The investigators measure the neck pain with Visual Analogue Scale (VAS) at the end of the intervention (through study completion, an average 11 days).
Cervical disability | Baseline.
  The investigators measure the cervical disability with Neck Disability Index (NDI) at baseline.
Cervical disability | Through study completion, an average 11 days.
  The investigators measure the cervical disability with Neck Disability Index (NDI) at the end of the intervention (through study completion, an average 11 days).
Motor control | Baseline.
  The investigators measure the motor control with Craniocervical Flexion Test (CCFT) at baseline.
Motor control | Through study completion, an average 11 days.
  The investigators measure the motor control with Craniocervical Flexion Test (CCFT) at the end of the intervention (through study completion, an average 11 days).

SECONDARY OUTCOMES:
Neck range of motion | Baseline.
  The investigators measure the neck range of motion with an inclinometer at baseline.
Neck range of motion | Through study completion, an average 11 days.
  The investigators measure the neck range of motion with an inclinometer at the end of the intervention (through study completion, an average 11 days).
Pressure pain threshold | Baseline.
  The investigators measure the pressure pain threshold with a digital algometer at baseline.
Pressure pain threshold | Through study completion, an average 11 days.
  The investigators measure the pressure pain threshold with a digital algometer at the end of the intervention (through study completion, an average 11 days).
Kinesiophobia | Baseline.
  The investigators measure the kinesiophobia with Tampa Scale for Kinesiophobia (TSK-11) at baseline.
Kinesiophobia | Through study completion, an average 11 days.
  The investigators measure the kinesiophobia with Tampa Scale for Kinesiophobia (TSK-11) at the end of the intervention (through study completion, an average 11 days).
Pain catastrophism | Baseline.
  The investigators measure the pain catastrophism with the Pain Catastrophizing Scale (PCS) at baseline.
Pain catastrophism | Through study completion, an average 11 days.
  The investigators measure the pain catastrophism with the Pain Catastrophizing Scale (PCS) at the end of intervention (through study completion, an average 11 days).
Anxiety and depression | Baseline.
  The investigators measure the anxiety and depression with the Hospital Anxiety and Depression Scale (HADS) at baseline.
Anxiety and depression | Through study completion, an average 11 days.
  The investigators measure the anxiety and depression with the Hospital Anxiety and Depression Scale (HADS) at the end of intervention (through study completion, an average 11 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Fisioterapia, Universidad de Valladolid, Soria, Spain